CLINICAL TRIAL: NCT03101995
Title: A Phase II Clinical Trial to Evaluate the Potential of Concomitant Chemoradiotherapy With Gemcitabine in Patients With Locally Advanced Carcinoma of Cervix and Renal Disease
Brief Title: Assessment of Gemcitabine as Chemoradiotherapy in Patients With Locally Advanced Carcinoma of Cervix and Renal Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: Instituto Nacional de Cardiologia Ignacio Chavez (Other); Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Lucely Cetina Pérez, MD, Master of Science, National Institute of Cancerología
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NationalIC; INCAN (Other: Instituto Nacional de Cancerología)
Record Dates: First submitted 2016-12-15; First posted 2017-04-05 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancer
Keywords: Treatment; Locally advanced cervical cancer; Renal failure; Gemcitabine
MeSH Terms: conditions — Uterine Cervical Neoplasms; Renal Insufficiency | interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: Phase II open, single arm, national, non-randomized clinical trial; to evaluate safety of gemcitabine in patients with locally advanced cervical cancer and renal dysfunction, referring to the INCAN.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gemcitabine (Experimental): Gemcitabine doses: 300 mg/m2/week for 6 weeks.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 300 mg/m2, prepared in 0.5 liters of sodium chloride 0.9%, IV administered in 30 minutes weekly for a maximum of 6 weeks.
  Radiotherapy will start the first week, or as soon as the blood count is normal or the patient has recovered after blood transfusion. Radiotherapy will be applied, using an external beam releasing 40-50.4 Gy in 20-28 fractions: 1.8 Gy/day for 5 days/week, during 4 to 6 weeks.
  Intracavitary brachytherapy will be added to reach a total EQD2 dosage (α/β=10) of 78-86 Gy.
  Other Names: Gemzar

SUMMARY:
From the global burden of Cervical Cancer (CC), 85% occurs in developing countries, representing 12% of cancer in women. In Mexico CC ranks second in incidence and mortality among women. The National Institute of Cancer in Mexico (lNCAN) receives annually about 500 patients with CC, 80% of which are diagnosed with locally advanced disease. Furthermore, 10 to 20% of these present kidney deterioration. The main reason for kidney disease is ureteral obstruction, other causes include age and comorbidities, such as diabetes and hypertension. The standard treatment for locally advanced disease consists in concomitant chemo-radiotherapy based on cisplatin (QT-RT), followed by brachytherapy, with an absolute benefit of 10%. However, the use of cisplatin in patients with renal disease may be questionable, considering it is a nephrotoxic treatment. Given that renal dysfunction limits the standard treatment efficiency because of the widely known nephrotoxicity of cisplatin, in most Cancer Centers of our country, patients with renal dysfunction receive only radiation therapy, even though it has proven less effective than concomitant QT-RT, limiting disease-free and overall survival of these patients. Venook et al. used gemcitabine as a radiosensitizer in patients with cancer and renal dysfunction. Our group, has observed encouraging results using gemcitabine as an alternative to cisplatin in concomitant treatment with radiotherapy, in CC patients with renal insufficiency. 89% of patients had complete response and improvement in renal function, with an enhanced creatinine clearance after treatment. Therefore, it is necessary to explore the safety of gemcitabine as an alternative treatment for CC patients with locally advanced disease and renal deterioration. We propose this clinical trial to assess the safety of treatment with gemcitabine and specifically on renal function in patients with renal deterioration. It is important to take into consideration that CC in advanced stages produces pain, transvaginal fetid discharge and general discomfort. It also causes side effects secondary to renal failure such as nausea, vomiting, fatigue, anemia, among others. These effects have a significant impact on the quality of life of these patients. Cancer treatment and its side effects, besides the implications of a nephrostomy catheter or ileostomy bag, determine the deterioration in the quality of life of the patient, during and sometimes after treatment. Thus it is of utmost importance to evaluate the factors that could help improve the quality of life of patients and explore the factors that deteriorate it. This clinical trial aims to generate scientific evidence to help make the best decisions concerning the treatment of patients with cervical cancer and renal impairment, and the impact on their quality of life.

DETAILED DESCRIPTION:
In Mexico, cervical cancer (CC) is the second most frequent cause of death among women, with a mortality rate of 4000 women/year. Concerning the treatment of these patients, there is evidence about the benefit of addition of chemotherapy to radiotherapy in patients with locally advanced CC, with an absolute benefit of 10% in overall survival and a significant reduction in local recurrence. Cisplatin is currently the standard treatment for CC. Evidence supports that the benefit of chemotherapy is achieved in those patients who receive at least 3 cycles of cisplatin at a dosage of 40mg/m2 weekly. The side effects of cisplatin include nephrotoxicity, neurotoxicity, nausea and vomiting, ototoxicity, electrolyte disturbance, and hemolytic anemia. For this reason, the choice of using cisplatin as a radiosensitizer requires careful consideration of the renal function of the patient, prior to the initiation of treatment. The glomerular filtration rate deteriorates with age and many patients have comorbid medical illnesses that further compromise the kidney. Gemcitabine has been tested as a single agent in CC for its radiosensitizing properties. Clinical profit has been reported along with reasonable tolerance to gemcitabine during radiotherapy. So it can be considered a good alternative treatment for the management of patients with ureteral obstruction and possible renal failure. Even though gemcitabine is well tolerated, the dosage for these patients should be considered with caution, since a specific dosage has not yet been recommended for cancer patients with renal dysfunction.

Our aim is to evaluate the safety of chemo-radiotherapy (QT-RT) concomitant with gemcitabine in patients with locally advanced cervical cancer IB2-IVA and renal deterioration. Our particular objectives are the following:

1. Evaluate the renal function before, during and after treatment with QT-RT concomitant with gemcitabine.
2. Assess the safety of concomitant QT-RT with gemcitabine, according to the common toxicity criteria in CTCEA v4.0.
3. Determine the objective and clinical response rate after treatment with QT-RT concomitant with gemcitabine.
4. Determine the incidence of percutaneous nephrostomy procedure.
5. Evaluate the clinical and cabinet criteria established by the protocol for the application of percutaneous nephrostomy or double J catheter and its impact on renal function.
6. Evaluate the patients' quality of life.
7. Determine the frequency of complications during and after treatment with QT-RT concomitant with gemcitabine.

Our aim is based on the following hypothesis. Patients with locally advanced CC IB2-IVA and renal dysfunction, that receive concomitant QT-RT with gemcitabine, tolerate the combination with a glomerular filtration rate of >60ml/min/1.73m2, show limited toxicity (Grade l-lll) and a response rate of at least 70%.

Methods.

Study design. It is a Phase II clinical trial, open, single-arm, national, nonrandomized, single-center; to evaluate the safety of gemcitabine in patients with locally advanced CC (IB2-IVA) and renal dysfunction, referring to the National Institute of Cancer in Mexico (INCAN). 18 patients will be included, with cervical malignant tumors of epithelial origin in the neck of the uterus, with renal impairment; candidates for QT-RT. Recruitment of patients will be performed in the first 12 months, with a follow up of 12 months, including 3 patients per month, to complete the total sample in one year (2017-2018).

Treatment. Based on treatment evidence the best dosage of gemcitabine in patients with adequate renal function is 300 mg/m2, prepared in 0.5 liters of sodium chloride 0.9%, IV administered in 30 minutes weekly for a maximum of 6 weeks, starting in the first week of radiotherapy or as soon as the blood count has recovered after blood transfusion. In our study design, patients will receive concomitant radiotherapy using an external beam releasing 40-50.4 Gy in 20-28 fractions: 1.8 Gy/day for 5 days/week, during 4 to 6 weeks. Intracavitary brachytherapy will be added to reach a total EQD2 dosage (α/β=10) of 78-86 Gy. In case retroperitoneal or para-aortic lymphnodes appear, patients will be treated with extended fields of radiotherapy at conventional doses. Dose will be adjusted up to 75% of the complete dosage in case of grade 3 (G3) leucopenia, G3 neutropenia, G3 thrombocytopenia, G3 diarrhea, radioepithelitis, or other G3 non hematological toxicity.

In case toxicity is not resolved within a week, treatment application may be delayed up to two weeks. If toxicity persists, subsequent doses will be suspended and the patient will receive only radiation therapy. Acute toxicity will be evaluated according to CTCAE (v. 4.03) toxicity criteria. When possible, chemotherapy treatment will coincide with radiotherapy. We will make every reasonable effort to ensure that radiotherapy treatment continues without interruption. Use of colony stimulating factor is allowed at the discretion of the researcher, it should not be administered within 24 hours prior or after treatment with chemotherapy. During each cycle, in all cases, creatinine clearance will be measured.

When an anaphylaxis or hypersensitivity reaction is suspected, gemcitabine infusion will be immediately stopped and replaced by saline solution. A physical examination including vital signs will be performed every 15 minutes, until the the patient's condition improves. Airways will be kept free. If a local reaction occurs (hives and angioneurotic edema), epinephrine and diphenhydramine should be administered. In case of bronchospasm, epinephrine, diphenhydramine, hydrocortisone, methylprednisolone and oxygen will be administered. In case of fever, antipyretic maneuvers will be performed and if the patient presents trembling, dipyrone will be administered. Emergency treatment will be evaluated and individualized by the immediate attention medic, who will administer the treatment that he deems pertinent to stabilize the patient.

The administration of other drugs will be performed if the physician considers it appropriate, however patients will not receive any other anti-cancer therapy under research, while participating in this study.

Sample size calculation. A sample space of 18 patients will be included if prior consent is acquired and if they meet the inclusion criteria.

This study will consider patient replacement in the following situation: if an adverse event occurs that prevents the patient to start the treatment previously described in the protocol after she has signed the informed consent.

Statistical analysis. A univariate analysis will be performed to describe the study population. Descriptive statistics will be used to obtain measures of central tendency and dispersion, as well as frequency of distribution for qualitative variables. A Bivariate analysis will be performed to observe the influence among variables. Kruskal-Walliss test will be used to evaluate variables of interest for different time points, before, during and after treatment. To assess differences in clinical response, we will use Zarah Fisher's exact test for categorical variables, and Mann-Whitney U test for quantitative variables. All confidence intervals will be constructed with a confidence of 95% (α=0.05). The interpretation of the study results will be responsibility of researchers. An interim analysis and a final report are planned; the first analysis will be made once the first 17 patients are included, and the final analysis is planned at 12 months after the last patient is included. Data processing and analysis will be performed with the SPSS package (version 19.0®) for Microsoft.

Safety analysis. Safety will be assessed in all patients who have received at least one chemotherapy application. To determine the safety of gemcitabine the following will be evaluated: to assess the safety of renal function, glomerular filtration rate will be evaluated; to assess systemic safety, number of required blood transfusions, clinical adverse events (including laboratory abnormalities), severity of each adverse event according to the toxicity criteria of CTCEA version 4.0, complications presented, and chronic toxicity according to RTOG criteria (Acute Radiation Morbidity Scoring Criteria). These will be evaluated 3 months after completing concomitant QT/RT treatment, in follow-up visits.

Procedures.

* Patients inclusion. Patients may start treatment within 21 days after being enrolled in the study. During the first seven days prior to the inclusion of the patients in the study, clinical history, complete physical examination including vital signs, weight, and general condition according to the ECOG scale, will be performed. Laboratory data (hematic biometry, serum electrolytes, glucose, serum creatinine, BUN, arterial blood gas, liver function enzymes, general urine test, urine culture, creatinine clearance in 24 hours, pregnancy test and HIV), will be measured within the first 14 days, prior to inclusion. Serum Cystatin C and urine albumin will also be determined at the National Institute of Cardiology in Mexico, within 21 days prior to inclusion. Imaging studies (PET-CT) will be performed to assess the tumor. To evaluate renal function, a bilateral renal ultrasound and a renal gammagraphy will be performed within 28 days prior to inclusion in the study. Additionally, thorax radiography will be required. If the patient presents hydronephrosis G3-4, a double J stent will be used for continent diversion, or a percutaneous nephrostomy procedure, and the patient may start treatment within the first 24-48 hours. Patients who meet the selection criteria will be included in the study to start treatment. Before initiating QT-RT, quality of life questionnaires will be applied. To have a more accurate nephrological examination, the results of all the laboratory tests previously mentioned for each patient, will be initially evaluated by nephrologists from the National Institute of Cardiology and the National Institute of Nutrition in Mexico.
* Visits during the study. After signing the informed consent, the patient will be informed when she will begin participating in the study (screening visit). If the patient complies with the inclusion criteria, a total of 21 visits will be scheduled. Of these, 8 visits will be given during treatment (an initial visit, 6 visits for QT-RT, 2 to 5 visits for brachytherapy), and 8 follow-up visits.
* Monitoring. Patient visits after QT-RT will be every 3 months during the follow-up year. Laboratory tests will be performed every visit (hematic biometry, serum electrolytes, glucose, serum creatinine, BUN, liver function enzymes, and general urine test). In case of clinical suspicion of progression, image studies (PET-CT), bilateral renal ultrasound and creatinine clearance calculation will be requested. The information obtained during this period will be limited physical examination, performance status assessment (ECOG), weight, measurement of tumor lesions by imaging studies, and date of progression or recurrence. Late adverse events will be evaluated at each scheduled visit. EORTC QLQ-30 and QLQ Cx-24 questionnaires will be applied during follow-up every 3 months for the first two years, and every 6 months for the following 3 years.
* Sample collection. No tissue or additional blood samples will be obtained, other than the blood samples used as part of the routine clinical laboratory tests.
* Informed consent acquisition. In the first visit, the consent will be read and explained to the patient, clarifying the risks and benefits involved in the study. Two witnesses, independent from the study, will be present when the consent is read and explained to the patient. The patient will have the choice to not participate or withdraw from the study at any time, her decision will not affect the quality of care and treatment that the attending physician will provide. The researcher will be governed by the ethical principles established in the Helsinki Accord. The physician will adequately respond all the matters of interest to the patient.

Ethical considerations. The Research Committee and the Ethics Committee of the National Institute of Cancer in Mexico has approved the protocol and the informed consent document. The approval will be valid for one year with the possibility of re-approval. Authorization from the national regulatory authority, the Federal Commission for the Protection against Health Hazards (COFEPRIS), will be requested.

Patients participating in this study will be informed, through the informed consent, of all the details concerning this trial. The patients who agree to participate in the trial will express their willingness by signing the informed consent document, being clarified that they can leave the trial at any time, if they wish to do so.

Regulatory considerations. This study abides by the ethical principles established by the international community, in accordance to the Good Clinical Practices, the Nüremberg Code, the Helsinki Accord, the Statement of Compliance with International Conference on Harmonization Guidelines for Good Clinical Practice, and the Regulations of the General Law of Health in the matter of research for health.

ELIGIBILITY:
Inclusion criteria.

1. Patients who give their written consent to participate in the study.
2. Women, 18-70 years of age, considering the following criteria:

   • In women of childbearing age: i. Negative serum pregnancy test at baseline (14 days prior to the start of QT-RT).

   ii. The patient must accept the use of any contraceptive method approved by the attending physician during the study and 12 weeks after the end of treatment.

   • Postmenopausal women must meet at least one of the following parameters for eligibility: i. Prior bilateral oophorectomy ii. Age ≥ 60 years iii. Age < 60 years, with amenorrhea for at least 12 months and levels of follicle stimulating hormone and estradiol within postmenopausal parameters.
3. Diagnosed with CC IB2-IVA, with or without retroperitoneal lymph nodes (para-aortic), smaller than 2 cm.
4. With histologic confirmation of squamous carcinoma, adenosquamous carcinoma, adenocarcinoma or glassy cells carcinoma.
5. Without previous treatment and medically able to receive gemcitabine.
6. Disease measurable by CT and/or MRI according to RECIST (v1.1) criteria.
7. Functional status of 0-3 according to WHO criteria.
8. Renal dysfunction defined by glomerular filtration (GF) <60 ml/min/1.73m2 calculated by the CKD-EPI formula.
9. Normal hematologic and liver function, as defined by the following parameters:

   * Hemoglobin > 10g/L. (Transfusion prior to the treatment is allowed to reach this level of hemoglobin).
   * Leucocytes > 4000/mm3.
   * Platelets > 100,000/mm3.
   * Total Bilirubin ≤1.5 times the upper normal limit (UNL).
   * Transaminases < 1.5 times the UNL.
10. Normal PA chest radiograph.

Exclusion criteria.

1. Patients with prior or concomitant malignancy, except non-melanoma skin carcinoma.
2. Patients with diabetes and/or hypertension with retinopathy or albuminuria >300.
3. Patients with evidence of active TB infection.
4. Patients infected with Human Immunodeficiency Virus (HIV).
5. Patients with a history of Systemic Lupus Erythematosus and other rheumatologic diseases that cause kidney damage.
6. Patients with vesicovaginal or vesicorectal fistula at the time of diagnosis.
7. Patients with uncontrolled intercurrent diseases including active infections that contraindicate QT, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, decompensated diabetes, difficult control hypertension and psychiatric illness.
8. Concomitant treatment with other experimental drugs.
9. Social, family or geographical conditions that suggest a poor adherence to the study.

Study discontinuation criteria.

1. Evidence of disease progression, if the researcher considers that the patient would benefit more with other therapy.
2. At the request of the patient.
3. By unacceptable toxicity.
4. Pregnancy.

Violation of starting criteria. Criteria must be followed punctually. If a patient were inappropriately included, she must be discontinued from the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-01-16 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Glomerular Filtration Rate | During and every 3 months after completing concomitant QT/RT treatment, for the first two years, and every 6 months for the following 3 years.
  Safety of gemcitabine regarding renal function will be assessed through glomerular filtration rate.
  An improvement of 10 ml/min/1.73m2 as compared to basal glomerular rate is expected by the end of treatment.

SECONDARY OUTCOMES:
Toxicity of gemcitabine in patients with carcinoma of cervix and renal disease | During and every 3 months after completing concomitant QT/RT treatment, for the first two years, and every 6 months for the following 3 years.
  Toxicity will be evaluated according to the toxicity criteria of CTCEA v. 4.03. A toxicity index of <4 is expected during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lucely C Cetina, MD, M.Sc., Principal Investigator — National Institute of Cancerología
Locations (1):
- National Institute of Cancer, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Green JA, Kirwan JM, Tierney JF, Symonds P, Fresco L, Collingwood M, Williams CJ. Survival and recurrence after concomitant chemotherapy and radiotherapy for cancer of the uterine cervix: a systematic review and meta-analysis. Lancet. 2001 Sep 8;358(9284):781-6. doi: 10.1016/S0140-6736(01)05965-7. PMID 11564482
- [Background] Brown JM. Carbogen and nicotinamide: expectations too high? Radiother Oncol. 1992 Jun;24(2):75-6. doi: 10.1016/0167-8140(92)90281-x. No abstract available. PMID 1386679
- [Background] Zarba JJ, Jaremtchuk AV, Gonzalez Jazey P, Keropian M, Castagnino R, Mina C, Arroyo G; GETICS (Grupo de Estudio, Tratamiento e Investigacion del Cancer del Sur) Argentina. A phase I-II study of weekly cisplatin and gemcitabine with concurrent radiotherapy in locally advanced cervical carcinoma. Ann Oncol. 2003 Aug;14(8):1285-90. doi: 10.1093/annonc/mdg345. PMID 12881394
- [Background] Duenas-Gonzalez A, Lopez-Graniel C, Gonzalez A, Reyes M, Mota A, Munoz D, Solorza G, Hinojosa LM, Guadarrama R, Florentino R, Mohar A, Melendez J, Maldonado V, Chanona J, Robles E, De la Garza J. A phase II study of gemcitabine and cisplatin combination as induction chemotherapy for untreated locally advanced cervical carcinoma. Ann Oncol. 2001 Apr;12(4):541-7. doi: 10.1023/a:1011117617514. PMID 11398890
- [Background] Chang PY, Dai MS, Ho CL, Yao NS. Administration of gemcitabine and cisplatin in cancer patients with renal failure under hemodialysis. J BUON. 2013 Oct-Dec;18(4):1058-61. PMID 24344039
- [Background] Pattaranutaporn P, Thirapakawong C, Chansilpa Y, Therasakvichya S, Ieumwananontachai N, Thephamongkhol K. Phase II study of concurrent gemcitabine and radiotherapy in locally advanced stage IIIB cervical carcinoma. Gynecol Oncol. 2001 Jun;81(3):404-7. doi: 10.1006/gyno.2001.6197. PMID 11371129
- [Background] Bosch A, Frias Z, Valda GC. Prognostic significance of ureteral obstruction in carcinoma of the cervix uteri. Acta Radiol Ther Phys Biol. 1973 Feb;12(1):47-56. doi: 10.3109/02841867309131091. No abstract available. PMID 4725645
- [Background] Cetina L, Rivera L, Candelaria M, de la Garza J, Duenas-Gonzalez A. Chemoradiation with gemcitabine for cervical cancer in patients with renal failure. Anticancer Drugs. 2004 Sep;15(8):761-6. doi: 10.1097/00001813-200409000-00004. PMID 15494637
- [Background] Rose PG, Ali S, Whitney CW, Lanciano R, Stehman FB. Impact of hydronephrosis on outcome of stage IIIB cervical cancer patients with disease limited to the pelvis, treated with radiation and concurrent chemotherapy: a Gynecologic Oncology Group study. Gynecol Oncol. 2010 May;117(2):270-5. doi: 10.1016/j.ygyno.2010.01.045. Epub 2010 Feb 24. PMID 20181381
- [Background] Tomimaru Y, Eguchi H, Satoh T, Tomokuni A, Asaoka T, Wada H, Marubashi S, Ogawa K, Takehara T, Mori M, Doki Y, Nagano H. Feasibility of pre-operative chemoradiotherapy with gemcitabine to treat pancreatic cancer in patients with impaired renal function. Jpn J Clin Oncol. 2015 Apr;45(4):343-8. doi: 10.1093/jjco/hyu224. Epub 2015 Jan 14. PMID 25589454
- [Background] Venook AP, Egorin MJ, Rosner GL, Hollis D, Mani S, Hawkins M, Byrd J, Hohl R, Budman D, Meropol NJ, Ratain MJ. Phase I and pharmacokinetic trial of gemcitabine in patients with hepatic or renal dysfunction: Cancer and Leukemia Group B 9565. J Clin Oncol. 2000 Jul;18(14):2780-7. doi: 10.1200/JCO.2000.18.14.2780. PMID 10894879
- [Background] Tanji N, Fukumoto T, Miura N, Yanagihara Y, Shirato A, Azuma K, Miyauchi Y, Kikugawa T, Shimamoto K, Yokoyama M. Combined chemotherapy with gemcitabine and carboplatin for metastatic urothelial carcinomas in patients with high renal insufficiency. Int J Clin Oncol. 2013 Oct;18(5):910-5. doi: 10.1007/s10147-012-0466-9. Epub 2012 Aug 31. PMID 22936563
- [Background] Grigsby PW. Cervical cancer: combined modality therapy. Cancer J. 2001 Jul-Aug;7 Suppl 1:S47-50. PMID 11504285
- [Background] Zahra MA, Taylor A, Mould G, Coles C, Crawford R, Tan LT. Concurrent weekly cisplatin chemotherapy and radiotherapy in a haemodialysis patient with locally advanced cervix cancer. Clin Oncol (R Coll Radiol). 2008 Feb;20(1):6-11. doi: 10.1016/j.clon.2007.10.007. Epub 2008 Jan 11. PMID 18191389